CLINICAL TRIAL: NCT06865001
Title: The Effect of Graded Motor Imagery on Pain, Range of Motion, Kinesiophobia, Position Sense and Quality of Life in Shoulder Impingement Syndrome
Brief Title: Effect of Graded Motor Imagery in Impingement
Acronym: Impingement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Associate Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: motor imagenaryfor Inpingement
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Shoulder; Impingement Syndrome; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): For patients diagnosed with shoulder impingemet, graded motor imagery will be applied in addition to 15 sessions of conventional treatment.
  Interventions: Other: Conventional treatment; Other: Graded motor imagery
- Control (Other): Patients diagnosed with shoulder impingemet will receive 15 sessions of conventional treatment.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Conventional treatment — Ultrasound, hotpack and TENS will be applied to both control and study groups as physical therapy modality. Then 15 sessions of Codman exercises, normal range of motion exercises and stretching exercises will be applied to both groups.
Other: Graded motor imagery — Graded motor imagery consists of three stages:
  1. limb lateralization task
  2. an imaginary limb movement task (motor imagery) and
  3. mirror therapy. Each session will consist of 12-15 minutes and 3 sets, with 5 minutes between sessions to rest and relax the limb. The application is planned for 30 minutes.
  Arms: Intervention

SUMMARY:
Purpose: This randomized controlled trial aims to investigate the effects of Graded Motor Imagery (GMI) added to conventional physiotherapy in patients with Grade-2 shoulder impingement syndrome. The primary objectives are to evaluate the impact of GMI on pain intensity, range of motion, kinesiophobia, joint position sense, and quality of life. The hypotheses tested are:

H0: GMI combined with conventional therapy has no effect on the aforementioned outcomes.

H1: GMI combined with conventional therapy significantly improves these outcomes.

Methodology: The study will include 30 participants (15 control, 15 intervention) diagnosed with Grade-2 shoulder impingement, recruited from a tertiary hospital. Participants will be randomly allocated into two groups:

Control Group: Receives 15 sessions of conventional physiotherapy (ultrasound, TENS, hotpack, and therapeutic exercises).

Intervention Group: Receives conventional therapy plus GMI, which includes three phases: (1) lateralization training (identifying left/right limb images), (2) motor imagery (mental rehearsal of functional movements), and (3) mirror therapy (visual feedback via mirror).

Outcome measures include pain (Visual Analog Scale), range of motion (digital goniometer), joint position sense (mobile app-based assessment), kinesiophobia (Tampa Scale), upper extremity function (DASH questionnaire), and quality of life (SF-36). Pre- and post-intervention evaluations will be conducted.

DETAILED DESCRIPTION:
Purpose:

This study is designed as a randomized controlled trial to evaluate the effectiveness of Graded Motor Imagery (GMI) as an adjunct to conventional physiotherapy in patients diagnosed with Grade-2 shoulder impingement syndrome. The primary aim is to assess the impact of GMI on several key outcomes, including pain intensity, range of motion, kinesiophobia (fear of movement), joint position sense, and quality of life. The study is motivated by the need to explore innovative rehabilitation techniques that address both the physical and neurological aspects of shoulder impingement syndrome, particularly in cases where conventional treatments may not yield optimal results.

The study is guided by two hypotheses:

Null Hypothesis (H0): The addition of GMI to conventional physiotherapy has no significant effect on pain, range of motion, kinesiophobia, joint position sense, or quality of life in patients with Grade-2 shoulder impingement syndrome.

Alternative Hypothesis (H1): The addition of GMI to conventional physiotherapy significantly improves pain, range of motion, kinesiophobia, joint position sense, and quality of life in these patients.

Methodology:

The study will be conducted at a tertiary hospital, with a sample size of 30 participants (15 in the control group and 15 in the intervention group). Participants will be recruited from patients diagnosed with Grade-2 shoulder impingement syndrome who meet the inclusion criteria, which include being between 18-65 years old, having a confirmed diagnosis, and being willing to participate in the study. Exclusion criteria include a history of upper extremity surgery, acute infections, or chronic neurological, psychiatric, or orthopedic conditions that could interfere with the study.

Participants will be randomly assigned to one of two groups using a simple randomization method:

Control Group: This group will receive 15 sessions of conventional physiotherapy, which includes modalities such as ultrasound, TENS (transcutaneous electrical nerve stimulation), hotpack application, and therapeutic exercises targeting shoulder mobility, strength, and stability.

Intervention Group: In addition to the conventional physiotherapy, this group will undergo a structured GMI program. The GMI protocol consists of three progressive phases:

Lateralization Training: Participants will be shown images of limbs and asked to quickly identify whether they are left or right. This phase aims to improve the brain's ability to distinguish between the affected and unaffected limbs.

Motor Imagery: Participants will mentally rehearse specific functional movements (e.g., combing hair, reaching for a cup) without physically performing them. This phase activates the premotor and primary motor cortices, helping to rewire the brain's motor pathways.

Mirror Therapy: A mirror will be used to create a visual illusion of the affected limb moving normally by reflecting the unaffected limb. This phase provides visual feedback to the brain, promoting cortical reorganization and reducing pain perception.

Outcome Measures:

The study will evaluate the following outcomes before and after the intervention:

Pain Intensity: Measured using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst pain imaginable.

Range of Motion: Assessed using a digital goniometer to measure shoulder flexion, extension, abduction, and internal/external rotation.

Kinesiophobia: Evaluated using the Tampa Scale for Kinesiophobia, which measures fear of movement and re-injury.

Joint Position Sense: Assessed using a mobile app-based method, where participants will position their shoulder at specific angles with eyes closed, and deviations from the target angle will be recorded.

Quality of Life: Measured using the SF-36 Health Survey, which evaluates physical and mental health across eight domains.

Upper Extremity Function: Assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, which evaluates the impact of shoulder pathology on daily activities.

Statistical Analysis:

Data will be analyzed using IBM SPSS Statistics (Version 23.0). The Shapiro-Wilk test will be used to check for normal distribution of data. For normally distributed data, parametric tests such as paired t-tests (for within-group comparisons) and unpaired t-tests (for between-group comparisons) will be used. For non-normally distributed data, non-parametric tests such as the Wilcoxon signed-rank test (within-group) and Mann-Whitney U test (between-group) will be applied. The significance level will be set at p < 0.05.

Expected Contributions:

This study aims to provide high-quality evidence on the effectiveness of GMI as an adjunct to conventional physiotherapy in the treatment of Grade-2 shoulder impingement syndrome. By exploring the impact of GMI on both physical and neurological outcomes, the study seeks to contribute to the development of more comprehensive rehabilitation protocols that address the multifaceted nature of chronic shoulder pain and dysfunction. The findings may also offer insights into the potential of GMI for other chronic pain conditions, paving the way for further research in this area.

Conclusion:

This randomized controlled trial represents a significant step forward in understanding the role of GMI in the rehabilitation of shoulder impingement syndrome. By integrating conventional physiotherapy with advanced neurorehabilitation techniques, the study aims to improve patient outcomes and enhance the quality of life for individuals suffering from this debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65,
* Volunteering to participate in the study,
* Diagnosed with Grade-2 shoulder impingement.

Exclusion Criteria:

* Not volunteering to participate in the study,
* Having undergone upper extremity surgery,
* History of previous shoulder surgery, shoulder subluxation or dislocation,
* Any mental or sensory problems,
* Acute infection or chronic disease of neurological, psychiatric, orthopedic, cardiological, rheumatological, etc. origin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 weeks
  In this study, the severity of shoulder pain will be evaluated with the Visual Analogue Scale. According to the VAS, pain intensity is graded as "no pain" 0 points and "worst unbearable pain" 10 points (10 cm scale).
Range of motion | 3 weeks
  In the study, a digital goniometer, which has been validated and reliable, was used to objectively evaluate the normal range of motion of the shoulder. Normal range of motion of the shoulder will be evaluated by measuring the range of motion of shoulder flexion, extension, abduction, internal rotation and external rotation movements.
Joint position sense | 3 weeks
  In this study, using this mobile application, the patient will perform 50-70-90 and 110 degrees of shoulder flexion with eyes open. Then, the patient will be asked to position the arm at the same angles with the eyes closed. Then the degrees of deviation will be calculated.

SECONDARY OUTCOMES:
The Short Form-36 Quality of Life Questionnaire | 3 weeks
  The Short Form-36, frequently used to assess quality of life, will be used. SF-36 consists of eight subscales including physical function, physical role, emotional function, social function, general health, mental health, pain and wellness. Each subscale scores between 0-100, and the scale is directly proportional to quality of life. A score of 100 indicates the best health status and a score of 0 indicates the worst health status.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH): | 3 weeks
  The validity of this questionnaire has been reported to be high in studies on the shoulder, elbow and wrist in the literature. It consists of 30 questions assessing the degree of difficulty in performing different activities in which the upper extremity is used in daily life in the last 1 week (21 questions), symptoms consisting of pain, activity-related pain, numbness, joint stiffness and weakness (5 questions), and the effects of pathologies on social life, sleep, work and psychological status (4 questions).
TAMPA Kinesiophobia Scale | 3 weeks
  It is a 17-question scale developed to measure fear of movement/reinjury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation,, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided